CLINICAL TRIAL: NCT03683173
Title: Multilevel Approaches for Promoting Physical Activity in Rural Communities
Brief Title: Promoting Physical Activity in Rural Communities
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Ross Brownson, Professor, Washington University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: R01CA211323 (NIH); R01CA211323 (NIH)
Record Dates: First submitted 2018-09-18; First posted 2018-09-25 (Actual); Results first posted 2024-01-08 (Actual); Last update posted 2024-01-08 (Actual); Status verified 2024-01

CONDITIONS: Physical Activity
Keywords: Physical Activity; Rural; Cancer Prevention
MeSH Terms: conditions — Motor Activity | interventions — Methods

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Multilevel Intervention (Experimental): Participants will receive the multilevel intervention consisting of community events, walking group formation, and short messaging service.
  Interventions: Behavioral: Intervention
- Control (No Intervention): Does not receive the multilevel intervention.

INTERVENTIONS:
Behavioral: Intervention — Participants in the intervention arm may receive community events, partake in walking groups, and receive short messaging service.
  Arms: Multilevel Intervention

SUMMARY:
The purpose of the study is to test a multilevel intervention's impact on increasing physical activity among rural residents. It is expected that participants who participate in more of the intervention (e.g., all levels) will increase their physical activity more than the control group and individuals who participate in less of the intervention (e.g., one level of the intervention).

DETAILED DESCRIPTION:
The study will test the independent and moderating effects of a multilevel intervention and the community environment on physical activity among rural residents. The multilevel intervention consists of community, interpersonal, and intrapersonal aspects. The community level intervention consists of community events. The interpersonal level intervention consists of walking group formation. The intrapersonal level intervention consists of cues provided by short message service messages (i.e., text messaging). A dose response relationship is expected in the intervention communities.

ELIGIBILITY:
Inclusion Criteria:

* Adults (18+)
* No cognitive impairments
* Able to physically active
* Willing to complete telephone survey at three time points
* Located in targeted communities in southeast Missouri

Exclusion Criteria:

* Participants not located in targeted communities

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1241 (Actual)
Dates: Start 2018-12-17 (Actual); Primary Completion 2022-12-24 (Actual); Study Completion 2022-12-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ross C Brownson, PhD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University in St. Louis, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Beck AM, Serrano N, Duncan D, Eyler AA, Gilbert A, Naghiloo F, Reis R, Tabak RG, Brownson RC. Cluster randomized multilevel intervention for promoting physical activity in rural communities. Front Public Health. 2025 Aug 29;13:1577056. doi: 10.3389/fpubh.2025.1577056. eCollection 2025. PMID 40951381
- [Derived] Serrano N, Beck A, Salvo D, Eyler A, Reis R, Steensma JT, Gilbert A, Brownson RC. Examining the Associations of and Interactions Between Intrapersonal and Perceived Environmental Factors With Objectively Assessed Physical Activity Among Rural Midwestern Adults, USA. Am J Health Promot. 2023 May;37(4):511-515. doi: 10.1177/08901171221134797. Epub 2022 Oct 21. PMID 36268648
- [Derived] Gilbert A, Beck A, Serrano N, Brownson RC. Objective Measures of Physical Activity in Rural Communities: Factors Associated With a Valid Wear and Lessons Learned. J Phys Act Health. 2022 Apr 1;19(4):267-274. doi: 10.1123/jpah.2021-0677. Epub 2022 Mar 10. PMID 35272263
- [Derived] Beck AM, Eyler AA, Aaron Hipp J, King AC, Tabak RG, Yan Y, Reis RS, Duncan DD, Gilbert AS, Serrano NH, Brownson RC. A multilevel approach for promoting physical activity in rural communities: a cluster randomized controlled trial. BMC Public Health. 2019 Jan 30;19(1):126. doi: 10.1186/s12889-019-6443-8. PMID 30700262

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 14 communities in southeastern Missouri were randomized to either the intervention group or the control group. Participants from these communities were consented and enrolled and the participant flow indicates the participants that started and completed the trial.
Units Other Than Participants: communities
Period: Enrolled and Completed Baseline Survey
Arm/Group | Multilevel Intervention | Control
Started | 627; 7 communities | 614; 7 communities
Completed | 627; 7 communities | 614; 7 communities
Not Completed | 0; 0 communities | 0; 0 communities
Period: Completed Follow-up
Arm/Group | Multilevel Intervention | Control
Started | 627; 7 communities | 614; 7 communities
Completed | 240; 7 communities | 238; 7 communities
Not Completed | 387; 0 communities | 376; 0 communities
Not completed — Unavailable | 235 | 217
Not completed — Refused | 69 | 59
Not completed — Disconnected phone | 65 | 95
Not completed — Health issue/deceased | 10 | 4
Not completed — Moved away | 8 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Multilevel Intervention | Control | Total
Number analyzed (Participants) | 627 | 614 | 1241
Age, Customized [Count of Participants; unit: Participants]
  <=18 years | 1 | 1 | 2
  Between 18 and 65 years | 406 | 393 | 799
  >65 years | 218 | 219 | 437
  Missing or Not Reported | 2 | 1 | 3
Sex/Gender, Customized [Count of Participants; unit: Participants] — This data is based on a question to the participant that asked "With what gender do you identify?"
  Participants
    Man | 202 | 197 | 399
    Woman | 424 | 417 | 841
    Refused | 1 | 0 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 11 | 9 | 20
  Not Hispanic or Latino | 615 | 604 | 1219
  Unknown or Not Reported | 1 | 1 | 2
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 521 | 512 | 1033
  Black or African American | 81 | 78 | 159
  American Indian/Alaska Native | 3 | 7 | 10
  Asian or Pacific Islander | 2 | 0 | 2
  Multi-racial | 18 | 10 | 28
  Not reported or missing | 2 | 7 | 9
Region of Enrollment [Number; unit: participants]
  United States | 627 | 614 | 1241
Household income before taxes [Count of Participants; unit: Participants]
  Less than $10,000 | 49 | 53 | 102
  $10,000 to under $15,000 | 46 | 48 | 94
  $15,000 to under $20,000 | 35 | 45 | 80
  $20,000 to under $25,000 | 43 | 36 | 79
  $25,000 to under $35,000 | 60 | 55 | 115
  $35,000 to under $50,000 | 77 | 78 | 155
  $50,000 to under $75,000 | 95 | 82 | 177
  $75,000 to under $100,000 | 53 | 71 | 124
  $100,000 to under $150,000 | 40 | 45 | 85
  $150,000 to under $200,000 | 9 | 5 | 14
  $200,000 or more | 16 | 14 | 30
  Missing or Not Reported | 104 | 82 | 186
Town [Count of Participants; unit: Participants] — Town that the participant reported living at the time of enrollment.
  Participants
    Piedmont | 56 | 0 | 56
    Doniphan | 0 | 93 | 93
    Perryville | 81 | 0 | 81
    Dexter | 0 | 56 | 56
    Poplar Bluff | 181 | 0 | 181
    Sikeston | 0 | 174 | 174
    Mountain View | 31 | 0 | 31
    Portageville | 0 | 30 | 30
    Kennett | 87 | 0 | 87
    West Plains | 0 | 124 | 124
    Charleston | 75 | 0 | 75
    Caruthersville | 0 | 61 | 61
    Jackson | 116 | 0 | 116
    Farmington | 0 | 76 | 76
Highest education level [Count of Participants; unit: Participants]
  Grades 1 - 8 (Elementary) | 7 | 15 | 22
  Grades 9 - 11 (Some High School) | 27 | 37 | 64
  Completed High School or GED equivalent | 168 | 161 | 329
  Some college or vocational program | 124 | 128 | 252
  Completed Associate degree (2-year program) | 91 | 69 | 160
  Completed Bachelors degree (4-year program) | 137 | 116 | 253
  Completed Masters degree | 53 | 59 | 112
  Beyond Masters degree | 20 | 27 | 47
  Missing or Not Reported | 0 | 2 | 2

OUTCOME MEASURES:

1. Primary Outcome: Change in Objective Physical Activity Measured by Accelerometer Measured at Baseline and 18-month Follow-up
Description: * Participants will wear an accelerometer to measure physical activity.
  * The outcome measure will measure the weekly minutes of moderate to vigorous physical activity.
  * Physical activity was measured using the Freedson Adult cutpoint categories from 1998. Each count was measured every 60 seconds/per minute.
    * Sedentary: 0-99 counts per minute
    * Light: 100-1951 counts per minute
    * Moderate: 1952-5724 counts per minute
    * Vigorous: 5725-9498 counts per minute
    * Very vigorous: 9499 and up counts per minute
Time Frame: Baseline and 18-month follow-up
Population: Only 56 participants (28 enrolled in the Multilevel Intervention Arm and 28 enrolled in the Control Arm) had valid data at baseline and at the 18-month follow-up.
Measure: Mean (Standard Deviation); unit: minutes per week
Arm/Group | Multilevel Intervention | Control
Number analyzed (Participants) | 28 | 28
minutes per week
  Baseline | 63.46 (84.58) | 96.94 (85.32)
  18-month follow-up | 74.02 (97.63) | 76.13 (72.79)

2. Secondary Outcome: Number of Participants Who Met the Subjective Physical Activity Recommendations as Measured by the Global Physical Activity Questionnaire at Baseline and 18-month Follow-up
Description: * Will use the Global Physical Activity Questionnaire to determine the number of participants who met the physical activity recommendations at baseline and at the 18-month follow-up.
  * The Global Physical Activity Questionnaire measures time spent in vigorous and moderate intensity physical activity in the domains of work, travel, and recreation. Participants will answer yes or no to their involvement in a given intensity (e.g., vigorous or moderate) in a given domain. If the participant answers 'yes' they will be asked on how many days do they partake in the activity, and for how many hours and/or minutes do they partake in the activity. A higher score equates to more physical activity. The range is from 0 minutes per week (no moderate physical activity in a week) to over 150 minutes per week (meeting recommendations) for moderate physical activity, and 0 minutes per week (no vigorous physical activity in a week) to over 75 minutes per week (meeting recommendations).
Time Frame: Baseline and 18-month follow-up.
Population: The number of participants analyzed includes only those who completed the questionnaire at the indicated time point.
Measure: Count of Participants; unit: Participants
Arm/Group | Multilevel Intervention | Control
Number analyzed (Participants) | 606 | 596
Participants
  Baseline | 292 | 287
  18-month follow-up: number analyzed (Participants) | 241 | 251
  18-month follow-up | 118 | 102

ADVERSE EVENTS:
Time Frame: Adverse events were followed from start of intervention or control through completion of 18-month follow-up.
Arm/Group | Multilevel Intervention | Control
All-Cause Mortality (participants affected / at risk) | 5/627 | 4/614
Serious Adverse Events (participants affected / at risk) | 0/627 | 0/614
Other Adverse Events (participants affected / at risk) | 0/627 | 0/614

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-10-26): https://cdn.clinicaltrials.gov/large-docs/73/NCT03683173/Prot_SAP_000.pdf